CLINICAL TRIAL: NCT00031551
Title: Evaluation of Efficacy and Mechanisms of an Anti-Inflammatory Intervention for Chemotherapy Related Mucosal Injury
Brief Title: Evaluation of Efficacy and Mechanisms of an Antiinflammatory Intervention for Chemotherapy Related Mucosal Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was not feasible to recruit required sample size from two clinical sites.
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 020133; 02-NR-0133 (Other: NIH CC)
Record Dates: First submitted 2002-03-07; First posted 2002-03-08 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Stomatitis
Keywords: Stomatitis; Oropharyngeal pain; TNF; Etanercept; Bone marrow transplantation; Chemotherapy; Cancer; Oral cavity; Oral mucous membranes; Randomized controlled clinical trial; Inflammation
MeSH Terms: conditions — Stomatitis; Neoplasms; Inflammation | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Main Study: Etanercept Mouthwash (Experimental): Etanercept 2.5 mg in 20cc mouthwash is swished and spit by the participant every 6 hours. The experimental mouthwash starts one day before conditioning chemotherapy is administered to the participant and continues until oral pain intensity and stomatitis severity scores are both 0, or by bone marrow transplant (BMT) Day +14, whichever occurs first.
  Interventions: Drug: Etanercept
- Main Study: Placebo Mouthwash (Placebo Comparator): Placebo 20cc mouthwash is swished and spit by the participant every 6 hours. The placebo mouthwash starts one day before conditioning chemotherapy is administered to the participant and continues until oral pain intensity and stomatitis severity scores are both 0, or by bone marrow transplant day (BMT) Day +14, whichever occurs first.
  Interventions: Drug: Placebo
- Pilot Study (No Intervention): Participants were enrolled in the pilot study to collect descriptive data about pain perception and laboratory techniques.

INTERVENTIONS:
Drug: Etanercept
  Other Names: Enbrel
  Arms: Main Study: Etanercept Mouthwash
Drug: Placebo
  Arms: Main Study: Placebo Mouthwash

SUMMARY:
This study consisted of two parts: the pilot study and the main study. The purpose of the pilot study is to demonstrate the effectiveness of planned laboratory techniques to assess for TNF-alpha gene expression from unstimulated saliva, plasma, and mucosal epithelial cells in patients who have chemotherapy-related stomatitis.

Main Study Description: Stomatitis is defined as inflammation of the mucous membranes of the oral cavity and oropharynx characterized by tissue erythema, edema, and atrophy, often progressing to ulceration. Stomatitis is a biologically complex, multifactorial, cancer treatment-related oral condition experienced by many oncology patients, which often leads to a cascade of negative sequelae including oropharyngeal pain, critical treatment alterations or cessation, and decreased quality of life. The optimal treatment strategies for stomatitis have not been established. There is a critical need to examine the pathogenesis of and to evaluate interventions for stomatitis and related acute oropharyngeal pain in the randomized controlled clinical trial setting using valid and reliable stomatitis assessment tools to both advance the science of cancer treatment-related oral toxicities and improve patient care. Therefore, the purpose of this randomized controlled clinical trial is to elucidate the role of inflammation in stomatitis by testing the effects of a novel tumor necrosis factor (TNF) fusion protein etanercept, (Enbrel, Immunex Corporation, Seattle, WA) on the incidence and severity of stomatitis. The actions of this fusion protein, which binds specifically to TNF preventing its interaction with cellular receptors and altering the inflammatory cascade, may provide insight into the role of inflammation in stomatitis. An etanercept effect is defined as a prevention or amelioration of stomatitis and acute oropharyngeal pain and/or changes in levels of tissue mediators. If stomatitis is primarily a consequence of a mucosal inflammatory response, then we hypothesize that this oral condition will be responsive to binding of TNF(alpha). Elaboration of the role of inflammatory cell signaling associated with stomatitis and the effect of TNF(alpha) may elucidate the mechanisms related to the pathogenesis of stomatitis and to other mucosal conditions.

Patients who are scheduled to receive autologous or allogenic peripheral blood stem cell or bone marrow transplant will be invited to participate in this study during a regularly scheduled pre-treatment visit. Written informed consent will be obtained from all participants. Patients will be randomized to receive either etanercept mouthwash or placebo, which will both be administered by protocol schedule. Stomatitis and oropharyngeal pain will be measured at baseline and at specified post-chemotherapy time points corresponding with the predicted stomatitis onset, peak, and healing time course. TNF(alpha) levels in buccal mucosa, analyzed by reverse transcriptase polymerase chain reaction techniques, and blood levels of pro-inflammatory cytokines, growth factors, and inflammatory mediators will also be measured at baseline and at specified post-chemotherapy time points corresponding with the predicted stomatitis onset, peak, and healing time course.

DETAILED DESCRIPTION:
This study consisted of two parts: the pilot study and the main study. The purpose of the pilot study is to demonstrate the effectiveness of planned laboratory techniques to assess for TNF-alpha gene expression from unstimulated saliva, plasma, and mucosal epithelial cells in patients who have chemotherapy-related stomatitis.

Main Study Description: Stomatitis is defined as inflammation of the mucous membranes of the oral cavity and oropharynx characterized by tissue erythema, edema, and atrophy, often progressing to ulceration. Stomatitis is a biologically complex, multifactorial, cancer treatment-related oral condition experienced by many oncology patients, which often leads to a cascade of negative sequelae including oropharyngeal pain, critical treatment alterations or cessation, and decreased quality of life. The optimal treatment strategies for stomatitis have not been established. There is a critical need to examine the pathogenesis of and to evaluate interventions for stomatitis and related acute oropharyngeal pain in the randomized controlled clinical trial setting using valid and reliable stomatitis assessment tools to both advance the science of cancer treatment-related oral toxicities and improve patient care. Therefore, the purpose of this randomized controlled clinical trial is to elucidate the role of inflammation in stomatitis by testing the effects of a novel tumor necrosis factor (TNF) fusion protein etanercept, (Enbrel) (Registered Trademark), Immunex Corporation, Seattle, WA) on the incidence and severity of stomatitis. The actions of this fusion protein, which binds specifically to TNF preventing its interaction with cellular receptors and altering the inflammatory cascade, may provide insight into the role of inflammation in stomatitis. An etanercept effect is defined as a prevention or amelioration of stomatitis and acute oropharyngeal pain and/or changes in levels of tissue mediators. If stomatitis is primarily a consequence of a mucosal inflammatory response, then we hypothesize that this oral condition will be responsive to binding of TNFa. Elaboration of the role of inflammatory cell signaling associated with stomatitis and the effect of TNFa may elucidate the mechanisms related to the pathogenesis of stomatitis and to other mucosal conditions.

Patients who are scheduled to receive autologous or allogeneic peripheral blood stem cell or bone marrow transplant will be invited to participate in this study during a regularly scheduled pre-treatment visit. Written informed consent will be obtained from all participants. Patients will be randomized to receive either etanercept 2.5mg in 20cc mouthwash or placebo 20cc mouthwash, which will both be administered by protocol schedule. Stomatitis and oropharyngeal pain will be measured at baseline and at specified post-chemotherapy time points corresponding with the predicted stomatitis onset, peak, and healing time course. TNFa levels in buccal mucosa, analyzed by real time polymerase chain reaction techniques, and blood levels of pro-inflammatory cytokines, growth factors, and inflammatory mediators will also be measured at baseline and at specified post-chemotherapy time points corresponding with the predicted stomatitis onset, peak, and healing time course.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female oncology patients who are enrolled in participating stomatogenic autologous or allogeneic PBSCT/BMT protocols, and are willing to participate in this study concurrently
  2. Able to understand and sign protocol consent or assent
  3. Age 16 years or older

EXCLUSION CRITERIA:

1. Pregnant or lactating females
2. Unable to follow oral rinsing directions
3. Intubation
4. Chronic use of medications confounding assessment of the inflammatory response (non-steroidal antiinflammatory drugs, antihistamines, and steroids- with the exception of decadron that is commonly used as an antiemetic in the PBSCT/BMT setting)
5. Pre-existing oral infection or upper respiratory infection that might maximize the possibility of an infection or sepsis contributing to a drug-related adverse event
6. Known hypersensitivity or allergic reaction to etanercept

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane M Fall-Dickson, PhD, Principal Investigator — National Institute of Nursing Research, National Institutes of Health
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Greenville Cancer Centers of the Carolinas, Greenville, South Carolina

REFERENCES:
- [Background] Seto BG, Kim M, Wolinsky L, Mito RS, Champlin R. Oral mucositis in patients undergoing bone marrow transplantation. Oral Surg Oral Med Oral Pathol. 1985 Nov;60(5):493-7. doi: 10.1016/0030-4220(85)90237-3. PMID 3903598
- [Background] Woo SB, Sonis ST, Monopoli MM, Sonis AL. A longitudinal study of oral ulcerative mucositis in bone marrow transplant recipients. Cancer. 1993 Sep 1;72(5):1612-7. doi: 10.1002/1097-0142(19930901)72:53.0.co;2-q. PMID 8348492
- [Background] Dose AM. The symptom experience of mucositis, stomatitis, and xerostomia. Semin Oncol Nurs. 1995 Nov;11(4):248-55. doi: 10.1016/s0749-2081(05)80005-1. PMID 8578032
- [Result] Fall-Dickson JM, Ramsay ES, Castro K, Woltz P, Sportes C. Oral mucositis-related oropharyngeal pain and correlative tumor necrosis factor-alpha expression in adult oncology patients undergoing hematopoietic stem cell transplantation. Clin Ther. 2007;29 Suppl:2547-61. doi: 10.1016/j.clinthera.2007.12.004. PMID 18164921
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-NR-0133.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study Participants: Participants were randomized to one of the following two interventions but the study was not unblinded.
  1. Etanercept 2.5 mg in 20cc mouthwash is swished and spit by the participant every 6 hours. The experimental mouthwash starts one day before conditioning chemotherapy is administered to the participant and continues until oral pain intensity and stomatitis severity scores are both 0, or by bone marrow transplant (BMT) Day +14, whichever occurs first.
  2. Placebo 20cc mouthwash is swished and spit by the participant every 6 hours. The placebo mouthwash starts one day before conditioning chemotherapy is administered to the participant and continues until oral pain intensity and stomatitis severity scores are both 0, or by bone marrow transplant day (BMT) Day +14, whichever occurs first.
Period: Overall Study
Arm/Group | Main Study Participants | Pilot Study
Started | 2 | 25
Completed | 0 | 25
Not Completed | 2 | 0
Not completed — Withdrew due to chemotherapy effects | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Participants | Pilot Study | Total
Number analyzed (Participants) | 2 | 25 | 27
Age, Continuous [Mean (Full Range); unit: years] | 59 [54 to 64] | 46 [32 to 68] | NA [NA to NA] — These numbers reflect two different populations in two different studies and were not analyzed together.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 13 | 13
  Male | 2 | 12 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2 | 16 | 18
  Hispanic | 0 | 6 | 6
  Black | 0 | 2 | 2
  Asian/Pacific Islander | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 25 | 27
Education [Number; unit: participants]
  Grade School | 0 | 2 | 2
  High School | 0 | 5 | 5
  Some College | 0 | 7 | 7
  College Graduate | 1 | 7 | 8
  Graduate School | 1 | 4 | 5
Cancer Diagnosis [Number; unit: participants]
  Breast Cancer | 0 | 7 | 7
  Non-Hodgkin's Lymphoma | 1 | 8 | 9
  Hodgkin's Lymphoma | 0 | 4 | 4
  Multiple Myeloma | 1 | 2 | 3
  Leukemia | 0 | 4 | 4
Cancer stage [Number; unit: participants]
  Stage II | 0 | 1 | 1
  Stage III | 1 | 13 | 14
  Stage IV | 0 | 5 | 5
  Unstaged | 0 | 1 | 1
  First Remission | 0 | 1 | 1
  Second Remission | 0 | 1 | 1
  Accelerated Phase | 0 | 1 | 1
  Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: What is the Clinical Efficacy of an Etanercept Mouthwash Used for the Treatment of Autologous or Allogeneic Peripheral Blood Stem Cell Transplant or Bone Marrow Transplant Treatment-related Stomatitis?
Description: Clinical efficacy will be determined by measurement of stomatitis grade and oropharyngeal pain.
Time Frame: 2 years
Population: Participants withdrew and analyses were terminated before any data collected.
Groups:
- Main Study: Etanercept Mouthwash: Etanercept 2.5 mg in 20cc mouthwash is swished and spit by the participant every 6 hours. The experimental mouthwash starts one day before conditioning chemotherapy is administered to the participant and continues until oral pain intensity and stomatitis severity scores are both 0, or by bone marrow transplant (BMT) Day +14, whichever occurs first.
  Etanercept
- Main Study: Placebo Mouthwash: Placebo 20cc mouthwash is swished and spit by the participant every 6 hours. The placebo mouthwash starts one day before conditioning chemotherapy is administered to the participant and continues until oral pain intensity and stomatitis severity scores are both 0, or by bone marrow transplant day (BMT) Day +14, whichever occurs first.
  Placebo
Arm/Group | Main Study: Etanercept Mouthwash | Main Study: Placebo Mouthwash
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: What is the Toxicity of an Etanercept Mouthwash Used for the Treatment of Autologous or Allogeneic Peripheral Blood Stem Cell Transplant or Bone Marrow Transplant Treatment -Related Stomatitis?
Description: Toxicity will be measured by the incidence of adverse events.
Time Frame: 2 years
Measure: Number; unit: event
Arm/Group | Main Study Participants
Number analyzed (Participants) | 2
event | 5

3. Other Pre Specified Outcome: Pilot Study: Mean Ratings of Oral Mucositis-related Oropharyngeal Pain Intensity on Day 9 (+/- 24 Hours) After Conditioning Chemotherapy (CT)
Description: Subjects rated pain using the Painometer, a hand-held tool with a visual analogue scale to rate overall pain intensity and a list of 14 sensory and 11 affective pain descriptors ranked by intensity values from 1 - 5. Subjects look at the list of sensory and affective words and select words that describe their pain, including Oral Pain and Oral Pain with Swallowing. . The weighted scores assigned to the words are added to obtain a pain intensity score for the sensory and the affective components. The overall pain intensity is measured on a visual analogue scale which has a range of 1 - 10 with high scores indicating higher pain intensity. The sensory and affective pain scores are otained by adding all of the respective intensity values. The range of possible sensory scores is from 0 - 48 and the range of possible affective scores is from 0 - 37. The sensory and affective scores may be added together to obtain the total pain intensity score, which may range from 0 - 85.
Time Frame: Day 9 (+/- 24 hours) after conditioning chemotherapy
Population: One subject was in critical condition at day 9 after CT, preventing data collection at this time
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pilot Study: Baseline Scores: Participants were enrolled in the pilot study to collect descriptive data about pain perception and laboratory techniques.
Arm/Group | Pilot Study: Baseline Scores | Pilot Study: Day 9 After CT Scores
Number analyzed (Participants) | 24 | 24
units on a scale
  Oral Pain: Overall pain intensity | 0.03 (0.16) | 1.38 (2.36)
  Oral Pain: Pain, Sensory Dimension | 0.12 (0.60) | 4.75 (11.58)
  Oral Pain: Pain, affective Dimension | 0.04 (0.20) | 3.33 (9.35)
  Oral Pain: Pain, Sensory and affective Dimensions | 0.16 (0.80) | 8.13 (19.79)
  Pain with Swallowing: Overall pain intensity | 0.03 (0.16) | 2.28 (3.38)
  Pain with Swallowing: Pain, Sensory Dimension | 0.08 (0.40) | 5.48 (11.69)
  Pain with Swallowing: Pain, Affective Dimension | 0 (0) | 4.09 (10.25)
  Pain with Swallowing:Sensory & Affective Dimension | 0.08 (0.40) | 9.61 (21.71)

4. Other Pre Specified Outcome: Pilot Study: Percentage of Participants Using Word Descriptors of Sensory and Affective Pain Selected by Subjects on Day 9 (+/- 24 Hours) After Conditioning Chemotherapy
Description: Participants selected from 14 word descriptors of sensory (S) pain and 11 word descriptors of affective (A) pain.
Time Frame: day 9 (+/- 24 hours) after conditioning chemotherapy
Population: One subject was in critical condition at day 9 after CT, preventing data collection at this time
Measure: Number; unit: percentage of participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 24
percentage of participants
  Sensory words: Cramping, radiation, sharp | 4.2
  Sensory: Splitting, shooting, stabbing, tearing | 8.3
  Sensory words: Dull, burning, crushing, pressing | 12.5
  Sensory words: Aching | 16.7
  Sensory words: Hurting | 20.8
  Sensory words: Sore | 29.2
  Sensory words: torturing, splitting, crushing | 4.2
  S:Cramping, shooting, radiating, stabbing, tearing | 8.3
  Sensory words: Dull, aching, pressing | 12.5
  Sensory words: Hurting Group 2 | 16.7
  Sensory words: Burning, sharp | 20.8
  Sensory words: Sore Group 2 | 29.2
  Affective words: Terrifying, torturing | 4.2
  Affective: Killing, tiring, unbearable, sickening | 8.3
  A: Nagging, agonizing, troublesome, miserable | 12.5
  Affective words: Annoying | 25.0
  Affective words: Torturing | 4.2
  Affective words: Killing, unbearable, terrifying | 8.3
  A: Agonizing, troublesome, tiring, sickening | 12.5
  Affective words: Miserable, nagging | 16.7
  Affective words: Annoying Group 2 | 20.8

ADVERSE EVENTS:
Description: Adverse events were not assessed for the pilot study.
Arm/Group | Main Study Participants | Pilot Study
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Participants (N=2) | Pilot Study (N=0)
Nausea (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes